CLINICAL TRIAL: NCT04018170
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, Phase I Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of JW1601
Brief Title: Single and Multiple Ascending Dose Study of JW1601 for Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JWP-FRC-101
Record Dates: First submitted 2019-03-25; First posted 2019-07-12 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JW1601 (Experimental): tablet formulation
  Interventions: Drug: Study drug
- Placebo (Placebo Comparator): tablet formulation identified with JW1601
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Study drug — oral administration, once daily. The doses will be ascending per cohort from 10 mg to 600 mg
  Other Names: JW1601
  Arms: JW1601
Drug: Placebo — oral administration, once daily. The matching placebo doses will be ascending per cohort from 1 to 4 tablets
  Arms: Placebo

SUMMARY:
This study is conducted to evaluate the safety/tolerability and PK/PD of JW1601 after oral administration in healthy Korean, Caucasian and Japanese adult volunteers

DETAILED DESCRIPTION:
This is a dose block-randomized, double-blind, placebo-controlled, single and multiple ascending dose study to assess the safety, tolerability and PK/PD profile by administering investigational product (IP) as a single dose (One time) or repeated doses (7 days, once a day) orally in a fasted state.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who have voluntarily given written informed consent to participate in the study and comply with all study requirements after getting detailed explanation and full understanding of the study

Exclusion Criteria:

- Subjects judged by the investigators unsuitable for participating in the study based on any other reasons

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after single ascending dose administration based on laboratory values, vital signs, ECG, physical examinations and Adverse Events monitoring | From Day 1 through Post Study Visit (Day 8)
  AE incidence and the value or the change from baseline such as vital signs, 12-lead ECG, and clinical laboratory tests will be compared by each group and placebo group.
Safety and tolerability in multiple ascending dose administration based on laboratory values, vital signs, ECG, physical examinations and Adverse Events monitoring | From Day 1 through Post Study Visit (Day 14)
  AE incidence and the value or the change from baseline such as vital signs, 12-lead ECG, and clinical laboratory tests will be compared by each group and placebo group.

SECONDARY OUTCOMES:
Cmax in plasma in single ascending dose administration | Baseline(Day 1) through Day 4
  Maximum concentration of drug in plasma
Tmax in plasma in single ascending dose administration | Baseline(Day 1) through Day 4
  Time to maximum plasma concentration
AUClast in plasma in single ascending dose administration | Baseline(Day 1) through Day 4
  Area under the plasma drug concentration-time curve to last measurement
Eosinophil shape change(%) in single ascending dose administration | Baseline(Day -1) through Day 4
  Imetit-induced eosinophil shape change
QT/QTc changes in single ascending dose administration | Baseline(Day -1), Day 1, Day 2
  12-lead ECG
C(max, ss) in plasma in multiple ascending dose administration | Baseline(Day 1) through Day 10
  Maximum concentration of drug in plasma (at steady state)
T(max,ss) in plasma in multiple ascending dose administration | Baseline(Day 1) through Day 10
  Time to maximum plasma concentration (at steady state)
AUC(τ,ss) in plasma in multiple ascending dose administration | Baseline(Day 1) through Day 10
  Area under the plasma drug concentration-time curve within a dosing interval(τ) at steady state
Eosinophil shape change(%) in multiple ascending dose administration | Baseline(Day -1) through Day 10
  Imetit-induced eosinophil shape change
QT/QTc changes in multiple ascending dose administration | Baseline(Day -1), Day 7, Day 8
  12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, MD, Principal Investigator — Severance Hospital
Locations (2):
- South Korea (2):
  - Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No